CLINICAL TRIAL: NCT04528147
Title: Yi Jin Jing Tiger Roaring Speech Rehabilitation With Real-Time Feedback Technique for Treatment of Speech Disorders in Parkinson's Disease: A Perspective Cohort Study
Brief Title: Yi Jin Jing Tiger Roaring Speech Rehabilitation With Real-Time Feedback Technique for PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Chief physician, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRS study
Record Dates: First submitted 2020-08-22; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Speech Disorders; Parkinson Disease
MeSH Terms: conditions — Speech Disorders; Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yi Jin Jing Tiger Roaring Speech Rehabilitation (Experimental): Yi Jin Jing tiger roaring speech rehabilitation with real-time feedback technique Duration: Each time requires an hour of training; Frequency: three times a week, 4 weeks in total.
  Interventions: Behavioral: Yi Jin Jing Tiger Roaring Speech Rehabilitation
- Conventional Speech Rehabilitation (Experimental): Patients will receive speech rehabilitation recommended by The Parkinson's Foundation.
  Duration: Each time requires an hour of training; Frequency: three times a week, 4 weeks in total.
  Interventions: Behavioral: Conventional Speech Rehabilitation

INTERVENTIONS:
Behavioral: Yi Jin Jing Tiger Roaring Speech Rehabilitation — A traditional Chinese medicine treatment
  Arms: Yi Jin Jing Tiger Roaring Speech Rehabilitation
Behavioral: Conventional Speech Rehabilitation — A active speech rehabilitation method recommended by the Parkinson's Foundation of America
  Arms: Conventional Speech Rehabilitation

SUMMARY:
Speech disorders affect more than 90% of patients with Parkinson's disease (PD). Neither of conventional drugs nor surgery can effectively improve speech function. Western speech rehabilitation is effective for speech disorders, but the domestic use of those methods used is limited. Our preliminary results revealed that traditional Chinese Yi jin jing tiger roaring speech rehabilitation is effectively in the treatment of speech disorders in PD, however, high-quality clinical evidence is still scarce. In order to solve this problem, we will conduct a prospective cohort study to explore the effects of Yi Jin Jing tiger roaring speech rehabilitation with real-time feedback technique on speech disorders in PD patients. This study will help to establish a set of Chinese Medicine treatment and objective evaluation methods for PD speech disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease
* Native language is Chinese
* VHI-10 score more than 10
* informed consent

Exclusion Criteria:

* Previous or concurrent medical history affecting swallowing function (laryngeal diseases such as vocal nodules, gastroesophageal reflux, and laryngeal cancer).
* History of serious psychosis
* Diagnosed by the investigators that patients with severe cardiac, liver and kidney diseases, or other serious health conditions
* Dementia (A Mini-Mental State Examination (MMSE) score of < 24), inability to comprehend the experimental protocol or voluntarily provide informed consent
* Lack of cooperation
* Additional reasons for exclusion at the discretion of the clinical investigator

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Differences in Voice Handicap Index (VHI) between treatment conditions in the on- and off- medication states | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  The Voice Handicap Index is a self-administered instrument, comprising 30 items on voice-related dysfunction. VHI has a range of 0 (normal voice function) to 120 (severe voice dysfunction).

SECONDARY OUTCOMES:
Differences in voice parameters between treatment conditions in the on- and off- medication states | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Voice recording at a sampling rate of 44.1 kHz using 16-bit quantification will be conducted in a sound-treated room using a microphone and a digital voice recorder with a mouth-to-microphone distance of 15 cm. The recorded voices will then be used for a composit acoustic analysis.
Differences in Swallowing Disturbance Questionnaire (SDQ) scores between treatment conditions in the on- and off- medication states. | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Differences in Swallowing Disturbance Questionnaire (SDQ) scores between treatment conditions in the on- and off- medication states.
Differences in Burg Balance Scale (BBS) scores between two treatment conditions in the on- and off- medication states. | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Burg Balance Scale measures patients' static and dynamic balance abilities. BBS score has a range of 0 (severe balance problems) to 56 (no balance problems).
Differences in Water Swallow Test (WST) scores between treatment conditions in the on- and off- medication states. | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  The Water Swallow Test is frequently used in clinical practice as a functional assessment to detect dysphagia, with stage 1 indicating severe dysphagia and stage 6 indicating normal swallowing function.
Differences in Beck Depression Inventory (BDI) scores between Treatment conditions. | Baseline, 4 weeks
  Beck Depression Inventory is a self-administered Instrument, contains 21 self-report items. The items are scored as 0, 1, 2, or 3. The score range is 0 (no depression) to 63 (severe depression).
Differences in Beck Anxiety Inventory (BAI) scores between treatment conditions. | Baseline, 4 weeks
  The BAI is a rating scale used to evaluate the severity of anxiety symptoms. It contains 21 self-report items. The items are scored as 0, 1, 2, or 3. The score range is 0-63. A total score of 0-7 is considered minimal range, 8-15 is mild, 16-25 is moderate, and 26-63 is severe.
Differences in 8-item Parkinson's Disease Questionnaire (PDQ-8) scores between treatment conditions. | Baseline, 4 weeks
  8-item Parkinson's Disease Questionnaire is a 8-item health-related quality of life instrument for subjects with Parkinson's Disease, which has a score range of 0 (good life quality) to 32 (very bad life quality).

CONTACTS AND LOCATIONS:
Locations (1):
- Functional neurosurgery of Shanghai jiaotong university affiliated Ruijin hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No